CLINICAL TRIAL: NCT00809159
Title: Randomized, Placebo Controlled Double Blind, Multi-center Phase II Proof-of-concept Study to Assess the Efficacy of AIN457 in Patients With Moderate to Severe Ankylosing Spondylitis
Brief Title: Double Blind, Placebo Controlled Study to Assess Efficacy of AIN457 in Moderate to Severe Ankylosing Spondylitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: CAIN457A2209; 2008-002631-33
Record Dates: First submitted 2008-12-16; First posted 2008-12-17 (Estimated); Results first posted 2015-09-18 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-08

CONDITIONS: Ankylosing Spondylitis
Keywords: ankylosing spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- Part 1 - AIN457A 10 mg/kg (Experimental): AIN457A 10.0 mg/kg was administered intravenously as a single dose.
  Interventions: Biological: AIN457
- Part 1 - Placebo (Placebo Comparator): Placebo to AIN457A was administered intravenously as a single dose
  Interventions: Drug: Placebo
- Parts 1 and 2 - AIN457A 1.0 mg/kg (Experimental): AIN457A 1.0 mg/kg was administered intravenously as 2 doses 21 days apart, i.e. the first dose on day 1 and the second dose on day 22.
  Interventions: Biological: AIN457
- Part 1 and 2 - AIN457 0.1 mg/kg (Experimental): AIN457A 0.1 mg/kg was administered intravenously as 2 doses 21 days apart, i.e. the first dose on day 1 and the second dose on day 22.
  Interventions: Biological: AIN457
- Part 1 and 2 - AIN457 10 mg/kg (Experimental): AIN457A 10.0 mg/kg was administered intravenously as 2 doses 21 days apart, i.e. the first dose on day 1 and the second dose on day 22.
  Interventions: Biological: AIN457

INTERVENTIONS:
Biological: AIN457 — AIN457A is a fully human recombinant IgG1 antibody that targets and neutralizes IL-17A.
  Arms: Part 1 - AIN457A 10 mg/kg; Part 1 and 2 - AIN457 0.1 mg/kg; Part 1 and 2 - AIN457 10 mg/kg; Parts 1 and 2 - AIN457A 1.0 mg/kg
Drug: Placebo — Placebo to AIN457
  Arms: Part 1 - Placebo

SUMMARY:
Evaluate the safety, tolerability and pharmacokinetics of AIN457 when administered as treatment of moderate to severe ankylosing spondylitis (AS).

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate to severe AS fulfilling the modified New York criteria for a diagnosis of AS and whose disease was not controlled on NSAIDS (on at least one NSAID over a period of at least 3 months at maximum dose). Minimum disease activity for inclusion of patients was assessed based on the ASAS core set domains: back pain & nocturnal pain score ≥ 4 despite concurrent NSAID use, PLUS a BASDAI score ≥ 4. Elevated CRP or ESR was not mandatory for study inclusion
* No evidence of liver disease or liver injury as indicated by abnormal liver function tests such as serum glutamic oxaloacetic transaminase (SGOT/AST), serum glutamic pyruvic transaminase (SGPT/ALT), gamma glutamyl transpeptidase (GGT), alkaline phosphatase, or serum bilirubin. The investigator was guided by criteria as outlined under exclusion criteria

Exclusion Criteria:

* For patients who were previously treated with TNF blockers, the following washout periods were required for these patients to be eligible to participate in the trial:
* month washout period prior to baseline for alefacept
* month washout period prior to baseline for adalimumab and certolizumab
* month washout prior to baseline for etanercept or infliximab
* For patients who were previously treated with immunosuppressive agents other than MTX, SSZ, and systemic corticosteroids, a 1-month washout period prior to baseline was required. Immunosuppressive agents included but were not limited to cyclosporine, mycophenolate, tacrolimus, and 5-aminosalicylic acid (5-ASA). Prednisone had to be kept at a stable dose 4 weeks before baseline and throughout the study and not to exceed 10 mg/day.
* MTX had to be kept at a stable dose 4 weeks before baseline and throughout the study and not to exceed 25 mg/week.
* SSZ had to be kept at a stable dose 4 weeks before baseline and throughout the study.
* In case of previous leflunomide treatment, a wash-out with oral cholestyramine could be considered as an alternative wash-out procedure to increase the elimination of leflunomide. Based on the notion that cholestyramine reduces plasma levels of the active leflunomide metabolite by approximately 40% in 24 hours and by 49% in 48 hours, cholestyramine was to be given orally at a dose of 8 g t.i.d. daily for 10 days. The patient could then be dosed with study drug not earlier than 2 weeks after the start of the cholestyramine wash-out procedure.
* Patients who were on NSAIDs had to be kept at a stable dose 4 weeks prior to baseline and throughout the study.
* Positive human immunodeficient virus (HIV: ELISA and Western blot) test result, Hepatitis B surface antigen (HBsAg) or Hepatitis C test result. Any active systemic infection within the past 2 weeks including a positive chest X-ray.
* Current signs or symptoms of severe, progressive, or uncontrolled renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, cardiac, neurologic, cerebral, psychiatric, chronic inflammatory diseases with the exception of psoriatic arthritis or other disease which in the clinical judgment of the investigator would make the patient unsuitable for the trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-03; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (19):
- United States (9):
  - Novartis Investigative Site, Paradise Valley, Arizona
  - Novartis Investigative Site, Springfield, Illinois
  - Novartis Investigative Site, Oklahoma City, Oklahoma
  - Novartis Investigative Site, Duncansville, Pennsylvania
  - Novartis Investigative Site, North Charleston, South Carolina
  - Novartis Investigative Site, Jackson, Tennessee
  - Novartis Investigative Site, Knoxville, Tennessee
  - Novartis Investigative Site, Benbrook, Texas
  - Novartis Investigative Site, Spokane, Washington
- Germany (4):
  - Novartis Investigative Site, Berlin, State of Berlin
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Herne
  - Novartis Investigative Site, München
- Netherlands (3):
  - Novartis Investigative Site, Meerssen, KR
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Maastricht
- United Kingdom (3):
  - Novartis Investigative Site, Leeds
  - Novartis Investigative Site, Newcastle upon Tyne
  - Novartis Investigative Site, Oxford

REFERENCES:
- [Derived] Baraliakos X, Borah B, Braun J, Baeten D, Laurent D, Sieper J, Emery P, McInnes IB, van Laar JM, Wordsworth P, Wollenhaupt J, Kellner H, Colin L, Vandenhende F, Radford K, Hueber W. Long-term effects of secukinumab on MRI findings in relation to clinical efficacy in subjects with active ankylosing spondylitis: an observational study. Ann Rheum Dis. 2016 Feb;75(2):408-12. doi: 10.1136/annrheumdis-2015-207544. Epub 2015 Aug 6. PMID 26248638
- [Derived] Baeten D, Baraliakos X, Braun J, Sieper J, Emery P, van der Heijde D, McInnes I, van Laar JM, Landewe R, Wordsworth P, Wollenhaupt J, Kellner H, Paramarta J, Wei J, Brachat A, Bek S, Laurent D, Li Y, Wang YA, Bertolino AP, Gsteiger S, Wright AM, Hueber W. Anti-interleukin-17A monoclonal antibody secukinumab in treatment of ankylosing spondylitis: a randomised, double-blind, placebo-controlled trial. Lancet. 2013 Nov 23;382(9906):1705-13. doi: 10.1016/S0140-6736(13)61134-4. Epub 2013 Sep 13. PMID 24035250

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Part 1 of the study, patients received 2 infusions spaced three weeks apart of 10 mg/kg AIN457 or placebo, and in Part 2 of the study, patients received 2 infusions spaced three weeks apart of 0.1 mg/kg, 1.0 mg/kg or 10 mg/kg AIN457, respectively.
Pre-assignment Details: Part 1 participants were randomized 4:1 to receive AIN457A or placebo. Part 2, the randomization ratio was to be 2:2:1 for the three dose groups, 0.1 mg/kg, 1 mg/kg and 10 mg/kg. More subjects were randomized to the 0.1 and 1mg/kg dose groups as compared to the 10 mg/kg group, as 24 subjects were already randomized to the 10 mg/kg group in Part 1.
Groups:
- Parts 1 and 2 - AIN457A 10 mg/kg: AIN457A 10 mg/kg was administered intravenously as 2 doses 21 days apart, i.e. the first dose on day 1 and the second dose on day 22.
- Part 1 and 2 - AIN457 1.0 mg/kg: AIN457A 1.0 mg/kg was administered intravenously as 2 doses 21 days apart, i.e. the first dose on day 1 and the second dose on day 22
- Part 1 and 2 - Placebo: Placebo to AIN457A was administered intravenously as a single dose
Period: Part 1
Arm/Group | Part 1 - AIN457A 10 mg/kg | Part 1 - Placebo | Parts 1 and 2 - AIN457A 10 mg/kg | Part 1 and 2 - AIN457 1.0 mg/kg | Part 1 and 2 - AIN457 0.1 mg/kg | Part 1 and 2 - Placebo
Started | 24 | 6 | 0 | 0 | 0 | 0
PK Analysis Set | 24 | 6 | 0 | 0 | 0 | 0
PD Analysis Set | 23 | 6 | 0 | 0 | 0 | 0
Completed | 16 | 3 | 0 | 0 | 0 | 0
Not Completed | 8 | 3 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 1 | 0 | 0 | 0 | 0
Not completed — Unsatisfactory therapeutic effect | 3 | 1 | 0 | 0 | 0 | 0
Period: Part 1 and 2
Arm/Group | Part 1 - AIN457A 10 mg/kg | Part 1 - Placebo | Parts 1 and 2 - AIN457A 10 mg/kg | Part 1 and 2 - AIN457 1.0 mg/kg | Part 1 and 2 - AIN457 0.1 mg/kg | Part 1 and 2 - Placebo
Started | 0 | 0 | 30 | 12 | 12 | 6
PK Analysis Set | 0 | 0 | 30 | 12 | 12 | 6
PD Analysis Set | 0 | 0 | 28 | 12 | 12 | 6
Completed | 0 | 0 | 20 | 7 | 6 | 3
Not Completed | 0 | 0 | 10 | 5 | 6 | 3
Not completed — Unsatisfactory therapeutic effect | 0 | 0 | 4 | 3 | 5 | 1
Not completed — Administrative problems | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 4 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Parts 1 and 2 - AIN457A 10 mg/kg | Part 1 and 2 - AIN457 1.0 mg/kg | Part 1 and 2 - AIN457 0.1 mg/kg | Part 1 and 2 - Placebo | Total
Number analyzed (Participants) | 30 | 12 | 12 | 6 | 60
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.7 (9.69) | 47.2 (10.50) | 42.8 (9.17) | 45.0 (9.96) | 42.8 (9.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 6 | 4 | 1 | 22
  Male | 19 | 6 | 8 | 5 | 38

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved ASAS20 Response
Description: Clinical response to treatment was assessed according to ASAS20 criteria. ASAS20 responder had improvement of 20% or more and absolute improvement of at least 1 units (on a scale of 0 [least] to 10 [worst]) from Baseline in at least 3 of the following 4 domains, with absence of deterioration (worsening of at least 20% an absolute Worsening of at least 1 unit) in the potential remaining domain: Patient's Global Assessment of Disease Activity; Total Back Pain visual analog scale (VAS); Function (Bath Ankylosing Spondylitis Functional Index (BASFI)); and Inflammation (mean of 2 morning stiffness-related Bath Ankylosing Spondylitis Disease Activity Index [BASDAI] scores
Time Frame: 6 Weeks
Population: Pharmacodynamic Analysis set: All patients with a least one evaluable post-treatment PD measurement and no major protocol deviations with impact on PD data were included. One subjects was excluded from the PD set in the AIN457 10mg/kg Part 1 due to protocol deviation
Measure: Number; unit: Percentage
Arm/Group | Part 1 - AIN457A 10 mg/kg | Part 1 - Placebo
Number analyzed (Participants) | 23 | 6
Percentage | 59.2 | 24.5

2. Primary Outcome: Change in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) Score From Baseline to 6 Weeks After First Infusion in Part 2
Description: ASAS20 as described in Primary Outcome. ASAS40 responder had improvement of 40% or more and absolute improvement of at least 2 units (on a scale of 0 [least] to 10 [worst]) from Baseline in at least 3 of the following 4 domains, with no deterioration in the potential remaining domain: Patient's Global Assessment of Disease Activity; Total Back Pain visual analog scale (VAS); Function (Bath Ankylosing Spondylitis Functional Index (BASFI)); and Inflammation (mean of 2 morning stiffness-related Bath Ankylosing Spondylitis Disease Activity Index [BASDAI] scores). ASAS 5/6 responder had improvement of 20% or more) from Baseline in at least 5 of the following 6 domains: Patient's Global Assessment of Disease Activity; Total Back Pain visual analog scale (VAS); Function (BASFI); and Inflammation (mean of 2 morning stiffness-related Bath Ankylosing Spondylitis Disease Activity Index [BASDAI] scores); Spinal Mobility (BASFI); Acute phase reactant (CRP)
Time Frame: 6 Weeks
Population: Pharmacodynamic Analysis set: All patients with a least one evaluable post-treatment PD measurement and no major protocol deviations with impact on PD data were included. One subjects was excluded from the PD set in the AIN457 10mg/kg Part 2 due to the absence of available post-baseline PD measurements
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Parts 1 and 2 - AIN457A 10 mg/kg | Part 1 and 2 - AIN457 1.0 mg/kg | Part 1 and 2 - AIN457 0.1 mg/kg | Part 1 and 2 - Placebo
Number analyzed (Participants) | 26 | 11 | 11 | 3
Units on a scale | -1.87 [-2.691 to -1.051] | -2.0151 [-3.275 to -0.755] | -1.2002 [-2.514 to 0.113] | -1.0577 [-2.893 to 0.777]

3. Secondary Outcome: Number of Participants Who Achieved ASAS20, ASAS40, and ASAS 5/6 Over Time in Part 1
Description: ASAS20 responder had improvement of 40% or more and absolute improvement of at least 2 units (scale of 0 [least] to 10 [worst]) from Baseline in at least 3 of the following 4 domains, with no deterioration in the potential remaining domain: Patient's Global Assessment of Disease Activity; Total Back Pain visual analog scale (VAS); Function (Bath Ankylosing Spondylitis Functional Index (BASFI)); and Inflammation (mean of 2 morning stiffness-related Bath Ankylosing Spondylitis Disease Activity Index [BASDAI] scores). ASAS 5/6 responder had improvement of 20% or more) from Baseline in at least 5 of the following 6 domains: Patient's Global Assessment of Disease Activity; Total Back Pain visual analog scale (VAS); Function (Bath Ankylosing Spondylitis Functional Index (BASFI)); and Inflammation (mean of 2 morning stiffness-related Bath Ankylosing Spondylitis Disease Activity Index [BASDAI] scores); Spinal Mobility (BASFI); Acute phase reactant (CRP)
Time Frame: Day8,15,29,week 6, 8, 10, 12, 16, 20, 24, 28
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Part 1 - AIN457A 10 mg/kg | Part 1 - Placebo
Number analyzed (Participants) | 23 | 6
Participants
  ASAS20 at Day 8 | 9 | 2
  ASAS20 at Day 15 | 9 | 1
  ASAS20 at Day 29 | 11 | 0
  ASAS40 at Day 8 | 4 | 0
  ASAS40 at Day 15 | 4 | 0
  ASAS40 at Day 29 | 8 | 0
  ASAS 5/6 at Day 8 | 5 | 1
  ASAS 5/6 at Day 15 | 5 | 0
  ASAS 5/6 at Day 29 | 8 | 0
  ASAS20 at week 6 | 14 | 1
  ASAS20 at week 8 | 8 | 1
  ASAS20 at week 10 | 9 | 0
  ASAS20 at week 12 | 9 | 1
  ASAS20 at week 16 | 8 | 1
  ASAS20 at week 20 | 6 | 1
  ASAS20 at week 24 | 7 | 0
  ASAS20 at week 28 | 7 | 1
  ASAS40 at week 6 | 7 | 1
  ASAS40 at week 8 | 5 | 0
  ASAS40 at week 10 | 5 | 0
  ASAS40 at week 12 | 3 | 0
  ASAS40 at week 16 | 3 | 1
  ASAS40 at week 20 | 2 | 1
  ASAS40 at week 24 | 3 | 0
  ASAS40 at week 28 | 2 | 0
  ASAS 5/6 at week 6 | 8 | 0
  ASAS 5/6 at week 8 | 7 | 0
  ASAS 5/6 at week 10 | 6 | 0
  ASAS 5/6 at week 12 | 3 | 0
  ASAS 5/6 at week 16 | 4 | 0
  ASAS 5/6 at week 20 | 2 | 1
  ASAS 5/6 at week 24 | 3 | 0
  ASAS 5/6 at week 28 | 1 | 0

4. Secondary Outcome: Number of Participants Who Achieved ASAS20, ASAS40, and ASAS 5/6 in Part 1 and 2 Combined
Description: a Bayesian model was fitted to the ASAS20 , ASAS40 and ASAS 5/6 response rates on active and placebo treatments. A Bayesian analysis had been chosen to allow the direct incorporation into the analysis of information about placebo response rates from historical data
Time Frame: Day 8,15,29,week 6, 8, 10, 12, 16, 20, 24, 28
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Parts 1 and 2 - AIN457A 10 mg/kg | Part 1 and 2 - AIN457 1.0 mg/kg | Part 1 and 2 - AIN457 0.1 mg/kg | Part 1 and 2 - Placebo
Number analyzed (Participants) | 28 | 12 | 12 | 6
Participants
  ASAS20 at day 8 (n=28,12,12,6) | 12 | 3 | 6 | 2
  ASAS20 at day 15 (n=28,12,12,5) | 11 | 7 | 4 | 1
  ASAS20 at day 29 (n=28,12,11,6) | 14 | 6 | 4 | 0
  ASAS40 at day 8 (n=28,12,12,6) | 6 | 2 | 2 | 0
  ASAS40 at day 15 (n=28,12,12,5) | 5 | 3 | 3 | 0
  ASAS40 at day 29 (28,12,11,6) | 10 | 3 | 1 | 0
  ASAS 5/6 at day 8 (28,12,12,6) | 6 | 3 | 5 | 1
  ASAS 5/6 at day 15 (n=28,12,12,5) | 5 | 5 | 2 | 0
  ASAS 5/6 at day 29 (n=28,12,11,6) | 9 | 5 | 3 | 0
  ASAS20 at week 6 (n=27,11,11,6) | 16 | 4 | 3 | 1
  ASAS20 at week 8 (n=28,11,11,6) | 10 | 4 | 3 | 1
  ASAS20 at week 10 (n=27,11,10,6) | 11 | 5 | 2 | 0
  ASAS20 at week 12 (n=27,12,11,6) | 12 | 3 | 4 | 1
  ASAS20 at week 16 (n=28,12,11,6) | 9 | 5 | 3 | 1
  ASAS20 at week 20 (n=28,12,11,6) | 6 | 4 | 2 | 1
  ASAS20 at week 24 (n=28,12,11,6) | 7 | 2 | 1 | 0
  ASAS20 at week 28 (n=28,11,11,6) | 8 | 2 | 2 | 1
  ASAS40 at week 6 (n=27,11,11,6) | 8 | 2 | 3 | 1
  ASAS40 at week 8 (n=28,11,11,6) | 5 | 2 | 2 | 0
  ASAS40 at week 10 (28,11,11,6) | 5 | 2 | 1 | 0
  ASAS40 at week 12 (n=27,12,11,6) | 3 | 2 | 3 | 0
  ASAS40 at week 16 (n=28,12,11,6) | 3 | 3 | 2 | 1
  ASAS40 at week 20 (n=28,12,11,6) | 2 | 1 | 2 | 1
  ASAS40 at week 24 (n=28,12,11,6) | 3 | 1 | 1 | 0
  ASAS40 at week 28 (n=28,11,11,6) | 3 | 0 | 1 | 0
  ASAS 5/6 at week 6 (n=28,11,11,6) | 9 | 3 | 2 | 0
  ASAS 5/6 at week 8 (n=28,11,11,6) | 7 | 4 | 1 | 0
  ASAS 5/6 at week 10 (n=27,11,10,6) | 6 | 4 | 1 | 0
  ASAS 5/6 at week 12 (n=28,12,11,6) | 5 | 2 | 1 | 0
  ASAS 5/6 at week 16 (n=28,12,11,6) | 5 | 5 | 2 | 0
  ASAS 5/6 at week 20 (n=28,12,11,6) | 2 | 3 | 1 | 1
  ASAS 5/6 at week 24 (n=28,12,11,6) | 3 | 2 | 1 | 0
  ASAS 5/6 at week 28 (n=28,11,10,6) | 2 | 0 | 1 | 0

5. Secondary Outcome: Magnetic Resonance Imaging (MRI) Inflammatory Scores at Baseline, Week 6 in Part 1
Description: The study used MRI with fat-saturating techniques such as short tau inversion recovery (STIR) to look for the presence of bone marrow edema. The Berlin modification of ASspiMRI-a (ASspiMRI-a) scoring technique assesses inflammation in each of the 23 disc vertebral units (DVU), capturing edema and erosion. Scores for each DVU range from 0-3 (0=normal; 1=minor bone marrow edema (less than25% of DVU; 3=severe bone marrow edema (more that 50% of DVU). The composite score ranges from 0 to 69, with higher scores indicating more severe inflammation
Time Frame: Baseline, week 6, week 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Part 1 - AIN457A 10 mg/kg | Part 1 - Placebo
Number analyzed (Participants) | 22 | 5
Score
  Baseline (n=22,5) | 9.2 (8.87) | 20.6 (20.18)
  Week 6 (n=22,3) | 6.6 (6.56) | 21.0 (24.56)
  Week 28 (n=16,5) | 5.7 (6.20) | 19.0 (19.33)

6. Secondary Outcome: Pharmacokinetics (PK) of AIN457: Time to Reach the Maximum Concentration After Drug Administration (Tmax) in Part 1
Description: Serum samples were collected pre-dose 2, 3, 4 and 24 hours after initiation of the infusions (Days 1 and 22), Weeks 1, 2, 4, 6, 8, 12, 16, 20, 24 and end of study/Week 28.
Time Frame: Week 28
Population: Pharmacokinetic Analysis set: All patients with quantifiable PK measurements and no major protocol deviations with impact on PK data. Due to several discontinuations, the full set of PK parameters could not be obtained in all treated patients. Patients who received only one infusion and/or had a too short PK sampling period were excluded.
Measure: Median (Full Range); unit: Days
Arm/Group | Part 1 - AIN457A 10 mg/kg
Number analyzed (Participants) | 23
Days | 21.07 [0.083 to 21.9]

7. Secondary Outcome: Pharmacokinetics (PK) of AIN457: Time to Reach the Maximum Concentration After Drug Administration (Tmax) in Part 1 and 2
Description: as for outcome 6
Time Frame: Week 28
Population: as for outcome 6
Measure: Median (Full Range); unit: Days
Arm/Group | Parts 1 and 2 - AIN457A 10 mg/kg | Part 1 and 2 - AIN457 1.0 mg/kg | Part 1 and 2 - AIN457 0.1 mg/kg
Number analyzed (Participants) | 28 | 12 | 12
Days | 21.08 [0.083 to 22.2] | 21.08 [0.125 to 23.0] | 21.12 [19.1 to 22.1]

8. Secondary Outcome: PK of AIN457: Observed Maximum Serum Concentration Following Drug Administration (Cmax) in Part 1
Description: as for outcome 6
Time Frame: Week 28
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Part 1 - AIN457A 10 mg/kg
Number analyzed (Participants) | 23
ug/mL | 357.7 (87.74)

9. Secondary Outcome: PK of AIN457: Observed Maximum Serum Concentration Following Drug Administration (Cmax) in Part 1 and 2
Description: as for outcome 6
Time Frame: Week 28
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Parts 1 and 2 - AIN457A 10 mg/kg | Part 1 and 2 - AIN457 1.0 mg/kg | Part 1 and 2 - AIN457 0.1 mg/kg
Number analyzed (Participants) | 28 | 12 | 12
ug/mL | 363.9 (82.30) | 33.13 (9.828) | 5.509 (5.418)

10. Secondary Outcome: PK of AIN457: Area Under the Serum Concentration-time Cure From Time Zero to the Time of Last Quantifiable Concentration (AUClast), Area Under the Serum Concentration-time Curve From Time Zero to (AUCinf) in Part 1
Description: as for outcome 6
Time Frame: Week 28
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: day*ug/mL
Arm/Group | Part 1 - AIN457A 10 mg/kg
Number analyzed (Participants) | 20
day*ug/mL
  AUCinf | 10510 (3036)
  AUClast | 10310 (2869)

11. Secondary Outcome: PK of AIN457: Area Under the Serum Concentration-time Cure From Time Zero to the Time of Last Quantifiable Concentration (AUClast), Area Under the Serum Concentration-time Curve From Time Zero to (AUCinf) in Part 1 and 2
Description: as for outcome 6
Time Frame: Week 28
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: day*ug/mL
Arm/Group | Parts 1 and 2 - AIN457A 10 mg/kg | Part 1 and 2 - AIN457 1.0 mg/kg | Part 1 and 2 - AIN457 0.1 mg/kg
Number analyzed (Participants) | 25 | 11 | 11
day*ug/mL
  AUCinf | 10880 (2983) | 1025 (276.0) | 198.0 (195.5)
  AUClast | 10630 (2818) | 993.0 (279.5) | 187.7 (190.7)

12. Secondary Outcome: PK of AIN457: Systemic Clearance From Serum Following Intravenous Administration (CL) in Part 1
Description: as for outcome 6
Time Frame: Week 28
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Liters/day
Arm/Group | Part 1 - AIN457A 10 mg/kg
Number analyzed (Participants) | 20
Liters/day | 0.1594 (0.04998)

13. Secondary Outcome: PK of AIN457: Systemic Clearance From Serum Following Intravenous Administration (CL) in Part 1 and 2
Description: as for outcome 6
Time Frame: Week 28
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Liters/day
Arm/Group | Parts 1 and 2 - AIN457A 10 mg/kg | Part 1 and 2 - AIN457 1.0 mg/kg | Part 1 and 2 - AIN457 0.1 mg/kg
Number analyzed (Participants) | 25 | 11 | 11
Liters/day | 0.1571 (0.04734) | 0.1718 (0.04942) | 0.1182 (0.05474)

14. Secondary Outcome: PK of AIN457: Volume of Distribution During the Terminal Phase Following Intravenous Elimination (Vz) in Part 1
Description: as for outcome 6
Time Frame: Week 28
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Part 1 - AIN457A 10 mg/kg
Number analyzed (Participants) | 20
Liters | 6.121 (0.999)

15. Secondary Outcome: PK of AIN457: Volume of Distribution During the Terminal Phase Following Intravenous Elimination (Vz) in Part 1 and 2
Description: as for outcome 6
Time Frame: Week 28
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Parts 1 and 2 - AIN457A 10 mg/kg | Part 1 and 2 - AIN457 1.0 mg/kg | Part 1 and 2 - AIN457 0.1 mg/kg
Number analyzed (Participants) | 25 | 11 | 11
Liters | 6.055 (0.943) | 6.481 (1.701) | 5.827 (2.887)

16. Secondary Outcome: PK of AIN457: Terminal Elimination Half-life (T1/2) in Part 1
Description: as for outcome 6
Time Frame: Week 28
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: day
Arm/Group | Part 1 - AIN457A 10 mg/kg
Number analyzed (Participants) | 20
day | 27.95 (5.624)

17. Secondary Outcome: PK of AIN457: Terminal Elimination Half-life (T1/2) in Part 1 and 2
Description: as for outcome 6
Time Frame: Week 28
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: day
Arm/Group | Parts 1 and 2 - AIN457A 10 mg/kg | Part 1 and 2 - AIN457 1.0 mg/kg | Part 1 and 2 - AIN457 0.1 mg/kg
Number analyzed (Participants) | 25 | 11 | 11
day | 28.09 (5.994) | 27.32 (7.234) | 34.31 (6.656)

18. Secondary Outcome: Mean Change Bath Ankylosing Spondylitis Metrology Index (BASMI) Score in Part 1 and 2
Description: BASMI measures the range of motion based on five clinical measurements: 1) cervical rotation, 2) tragus to wall distance, 3) lumbar side flexion, 4) lumbar flexion (modified Schober's) and 5) intermalleolar distance. BASMI 0 = indicates mild disease involvement, 1 = moderate disease, and 2 = severe disease involvement. The results for cervical rotation and lumbar side flexion are the means of the left and right measurements. Scoring range 0-10. The higher the BASMI score, the more severe was the subject's limitation of movement
Time Frame: Baseline, day 8,15,29, week 6,8,10,12,16,20,24,28
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Parts 1 and 2 - AIN457A 10 mg/kg | Part 1 and 2 - AIN457 1.0 mg/kg | Part 1 and 2 - AIN457 0.1 mg/kg | Part 1 and 2 - Placebo
Number analyzed (Participants) | 28 | 12 | 12 | 6
Score
  Day 8 (n=28,12,12,5) | -0.121 (0.7969) | -0.117 (0.6293) | -0.233 (0.9335) | 0.240 (0.2966)
  Day 15 (n=28,12,12,5) | -0.200 (0.7364) | -0.383 (0.5937) | -0.350 (0.7775) | 0.160 (0.8764)
  Day 29 (n=28,12,11,6) | -0.157 (0.8404) | -0.417 (0.7259) | -0.382 (1.0713) | 0.100 (0.2098)
  Week 6 (n=27,11,11,3) | -0.281 (0.8138) | -0.436 (0.7256) | -0.291 (0.8961) | 0.133 (0.6110)
  Week 8 (n=26,11,11,3) | -0.238 (0.8100) | -0.518 (1.0925) | -0.509 (0.9523) | -0.133 (0.6110)
  Week 10 (n=25,11,10,3) | -0.376 (0.8686) | -0.200 (0.9077) | -0.400 (0.6325) | -0.067 (0.4163)
  Week 12 (n=25,12,11,3) | -0.384 (0.8887) | -0.267 (0.7738) | -0.455 (0.9883) | -0.200 (0.6928)
  Week 16 (n=24,10,8,3) | -0.200 (0.8299) | -0.400 (0.7424) | -0.550 (0.9304) | 0.400 (0.8000)
  Week 20 (n=21,9,6,3) | -0.143 (0.9168) | -0.356 (0.6064) | -0.633 (1.0912) | -0.200 (1.5875)
  Week 24 (n=20,8,5,3) | -0.250 (0.7564) | 0.200 (0.5657) | -0.800 (1.1045) | 0.400 (0.7211)
  Week 28 (n=28,11,11,5) | -0.036 (0.7345) | -0.182 (0.9527) | -0.230 (0.8145) | 0.400 (0.4690)

19. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) in Part 1 and 2
Description: The BASDAI consists of a 1 through 10 scale (1 being no problem and 10 being the worst problem), which was used to answer 6 questions pertaining to the 5 major symptoms of AS: Fatigue, Spinal pain, Joint pain / swelling, areas of localized tenderness (called enthesitis, or inflammation of insertion sites of tendons and ligaments), morning stiffness duration, and morning stiffness severity. The physician will globally assess the subject's current disease state using a visual analog scale (VAS) scale with 0 being very good and 100 being very bad.
Time Frame: Baseline, day 8,15,29,week 6,8,10,12,16,20,24,28
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Score
Arm/Group | Parts 1 and 2 - AIN457A 10 mg/kg | Part 1 and 2 - AIN457 1.0 mg/Kg | Part 1 and 2 - AIN457 0.1 mg/kg | Part 1 and 2 - Placebo
Number analyzed (Participants) | 28 | 12 | 12 | 6
Score
  Day 8 (n=28,12,11,6) | -1.7011 [-2.533 to -0.870] | -1.2793 [-2.559 to 0.001] | -1.2920 [-2.635 to 0.051] | -1.0837 [-2.737 to 0.570]
  Day 15 (n=28,12,11,5) | -1.7094 [-2.485 to -0.934] | -2.1256 [-3.317 to -0.934] | -1.1263 [-2.376 to 0.124] | -0.6417 [-2.199 to 0.915]
  Day 29 (n=28,12,11,6) | -2.2530 [-3.096 to -1.410] | -2.4237 [-3.722 to -1.126] | -1.3886 [-2.750 to -0.028] | -0.7839 [-2.464 to 0.896]
  Week 6 (n=26,11,11,3) | -1.8713 [-2.691 to -1.051] | -2.0151 [-3.275 to -0.755] | -1.2002 [-2.514 to 0.113] | -1.0577 [-2.893 to 0.777]
  Week 8 (n=26,11,11,3) | -1.3863 [-2.189 to -0.584] | -1.6994 [-2.933 to -0.466] | -1.2020 [-2.485 to 0.081] | -1.4619 [-3.401 to 0.477]
  Week 10 (n=24,11,9,3) | -1.6246 [-2.389 to -0.860] | -1.7402 [-2.909 to -0.571] | -1.0800 [-2.313 to 0.153] | -0.8527 [-2.558 to 0.853]
  Week 12 (n=24,12,11,3) | -1.4744 [-2.336 to -0.613] | -1.3755 [-2.688 to -0.063] | -1.6834 [-3.059 to -0.307] | -1.3529 [-3.354 to 0.648]
  Week 16 (n=24,10,8,3) | -1.3990 [-2.237 to -0.562] | -2.3081 [-3.589 to -1.027] | -1.7628 [-3.143 to -0.383] | -1.4083 [-3.415 to 0.598]
  Week 20 (n=21,9,6,3) | -1.2072 [-2.011 to -0.403] | -1.4070 [-2.632 to -0.183] | -1.1596 [-2.521 to 0.202] | -1.5864 [-3.385 to 0.212]
  Week 24 (n=20,8,5,3) | -1.1318 [-2.001 to -0.262] | -1.0035 [-2.343 to 0.336] | -0.8020 [-2.305 to 0.701] | -1.2048 [-3.201 to 0.792]
  Week 28 (n=28,11,11,5) | -0.7373 [-1.487 to 0.012] | -0.8980 [-2.057 to 0.261] | -1.2227 [-2.432 to -0.013] | -0.9722 [-2.526 to 0.582]

20. Secondary Outcome: Mean Change in Maastricht Ankylosing Spondylitis Enthesitis Score (MASES) in Part 1
Description: MASES is measured by scoring of entheses of 0 (no tenderness) to 3 (severe tenderness) at 13 sites on the body. The score was derived as the sum of the 13 scores divided by 3 and the total range is 0 (no tenderness) to 13 (severe tenderness).
Time Frame: Baseline, day 8,15,29,week, 6, 8,10,12,16,20,24,28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Part 1 - AIN457A 10 mg/kg | Part 1 - Placebo
Number analyzed (Participants) | 23 | 6
Score
  Day 8 (n=23,6) | -1.3 (2.46) | 0.7 (1.37)
  Day 15 (n=23,5) | -1.3 (2.53) | 2.4 (2.51)
  Day 29 (n=23,6) | -1.0 (2.80) | -0.3 (1.97)
  Week 6 (n=22,3) | -1.5 (3.10) | -0.3 (0.58)
  Week 8 (n=21,3) | -1.0 (2.77) | 0.0 (0.0)
  Week 10 (n=20,3) | -1.3 (3.24) | -0.3 (0.58)
  Week 12 (n=20,3) | -1.2 (3.09) | -0.3 (0.58)
  Week 16 (n=30,3) | -0.9 (3.69) | -0.3 (0.58)
  Week 20 (n=18,3) | 0.2 (3.55) | 0.3 (1.53)
  Week 24 (n=17,3) | -1.3 (2.11) | -0.3 (0.58)
  Week 28 (n=23,5) | -0.4 (3.86) | 1.2 (1.30)

21. Secondary Outcome: Mean Change in Maastricht Ankylosing Spondylitis Enthesitis Score (MASES) in Part 1 and 2
Description: as for outcome 20
Time Frame: Day 8,15,29,week, 6, 10,12,16,20,24,28
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Parts 1 and 2 - AIN457A 10 mg/kg | Part 1 and 2 - AIN457 1.0 mg/kg | Part 1 and 2 - AIN457 0.1 mg/kg | Part 1 and 2 - Placebo
Number analyzed (Participants) | 28 | 12 | 12 | 6
Score
  Day 8 (n=28,12,12,6) | -1.321 (2.7763) | -1.917 (2.2344) | -0.583 (1.0836) | 0.667 (1.3663)
  Day 15 (n=28,12,12,5) | -1.393 (2.7667) | -1.167 (1.9924) | -1.167 (1.9462) | 2.400 (2.5100)
  Day 29 (n=28,12,11,6) | -1.143 (2.9779) | -2.083 (2.2344) | -0.545 (0.6876) | -0.333 (1.9664)
  Week 6 (n=27,11,11,3) | -1.556 (3.2026) | -0.339 (3.1318) | -0.364 (1.0269) | -0.333 (0.5774)
  Week 8 (n=26,11,11,3) | -1.154 (2.9758) | -1.273 (1.6787) | 0.455 (2.2523) | 0.0 (0.0)
  Week 10 (n=25,11,10,3) | -1.360 (3.3277) | -1.091 (3.1450) | -0.800 (0.9189) | -0.333 (0.5774)
  Week 12 (n=25,12,11,3) | -1.280 (3.2342) | -1.167 (4.1304) | -0.636 (1.8040) | -0.333 (0.5774)
  Week 16 (n=24,10,8,3) | -1.042 (3.7819) | -0.600 (3.4705) | 0.500 (1.6903) | -0.333 (0.5774)
  Week 20 (n=21,9,6,3) | -0.238 (3.8458) | -0.333 (3.7749) | -0.667 (1.3663) | 0.333 (1.5275)
  Week 24 (n=20,8,5,3) | -1.400 (2.2572) | -1.000 (3.7417) | 0.600 (1.9494) | -0.333 (0.5774)

22. Secondary Outcome: Change From Baseline in the Health Related Quality of Life (HRQoL) by Using the SF-36 Physical Component, and the ASQoL (Ankylosing Spondylitis Quality of Life Instrument) in Part 1.
Description: The Short Form (36) Health Survey (SF-36) measures the impact of disease on overall quality of life and consists of eight subscales (physical function, pain, general and mental health, vitality, social function, physical and emotional health) which can be aggregated to derive a physical-component summary score and a mental-component summary score. Scores range for each subscale from 0 to 10, and the composite score ranges from 0 to 100, with higher scores indicative of better health. ASQoL determined subject's quality of life and is comprised of 18 questions (yes or no) to be completed by the subject. Each statement on the ASQoL is given a score of "1" or "0." All item scores were summed to give a total score or index. Total scores ranged from 0 (good quality of life) to 18 (poor quality of life) related to ability to cope, relationships, mood, sleep, motivation, activities of everyday living, independence, and social life. Decrease in ASQoL score represents improvement.
Time Frame: SF-36:Baseline, week 12, week 28; ASQoL: Baseline, Day 29, week 12, week 28
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Part 1 - AIN457A 10 mg/kg | Part 1 - Placebo
Number analyzed (Participants) | 23 | 6
Score
  Baseline SF36 Mental component (n= 22,6) | 38.71 (10.78) | 39.57 (14.63)
  Baseline SF36 physical component (n=22,6) | 31.42 (5.2) | 30.11 (6.71)
  Week 12 SF36 Mental component (n=20,3) | 43.45 (10.56) | 56.57 (5.39)
  Week 12 SF36 Physical component (n=20,3) | 32.84 (6.39) | 28.95 (1.8)
  Week 28 SF36 Mental component (n=21,4) | 41.65 (9.86) | 40.51 (15.22)
  Week 28 SF36 Physical component (n=21,4) | 32.2 (5.68) | 33.96 (8.73)
  Change from Baseline to Day 29 ASQoL (n=21,6) | -2.9 (4.04) | -0.7 (2.58)
  Change from Baseline to Week 12 ASQoL (n=18,3) | -2.3 (3.05) | 0.0 (1.00)
  Change from Baseline to Week 28 ASQoL (n=20,4) | -1.2 (3.71) | -1.3 (2.06)

23. Secondary Outcome: Change From Baseline in the Health Related Quality of Life (HRQoL) by Using the SF-36 Physical Component, and the ASQoL (Ankylosing Spondylitis Quality of Life Instrument) in Part 1 and 2.
Description: The SF-36 measures the impact of disease on overall quality of life and consists of eight subscales (physical function, pain, general and mental health, vitality, social function, physical and emotional health) which can be aggregated to derive a physical-component summary score and a mental-component summary score. ASQoL determined subject's quality of life and is comprised of 18 questions (yes or no) to be completed by the subject. Each statement on the ASQoL is given a score of "1" or "0." All item scores were summed to give a total score or index. Total scores ranged from 0 (good quality of life) to 18 (poor quality of life) related to ability to cope, relationships, mood, sleep, motivation, activities of everyday living, independence, and social life. Decrease in ASQoL score represents improvement.
Time Frame: SF-36: Baseline, week 12, week 28; ASQoL: Baseline, day 29, week 12, week 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Parts 1 and 2 - AIN457A 10 mg/kg | Part 1 and 2 - AIN457 1.0 mg/kg | Part 1 and 2 - AIN457 0.1 mg/kg | Part 1 and 2 - Placebo
Number analyzed (Participants) | 28 | 12 | 12 | 6
Score
  Baseline SF36 Mental component (n=27,12,12,6) | 38.97 (10.91) | 39.46 (11.95) | 51.9 (8.7) | 39.57 (14.63)
  Baseline SF36 Physical component (n=27,12,12,6) | 30.95 (6.34) | 26.17 (7.63) | 33.53 (7.47) | 30.11 (6.71)
  Week 12 SF36 Mental component (n=25,11,10,3) | 44.37 (11.05) | 38.45 (10.13) | 49.7 (11.74) | 56.57 (5.39)
  Week 12 SF36 Physical component (n=25,11,10,3) | 32.71 (6.24) | 31.3 (7.67) | 35.81 (5.29) | 28.05 (1.8)
  Week 28 SF36 Mental component (n=26,11,10,4) | 40.94 (10.56) | 36.6 (10.3) | 46.96 (9.67) | 40.51 (15.22)
  Week 28 SF36 Physical component (n=26,11,10,4) | 31.85 (5.3) | 29.95 (6.92) | 35.54 (5.9) | 33.96 (8.73)
  Change from Baseline to Day 29 ASQoL(n=26,11,10,6) | -3.2 (3.78) | -3.1 (2.63) | -0.7 (2.26) | -0.7 (2.58)
  Change from Baseline to Week 12 ASQoL(n=23,11,9,3) | -2.7 (2.91) | -2.7 (4.71) | -1.3 (3.16) | 0.0 (1.00)
  Change from Baseline to Week 28 ASQoL(n=25,11,9,4) | -1.4 (3.37) | -1.3 (3.66) | -0.9 (2.15) | -1.3 (2.06)

ADVERSE EVENTS:
Groups:
- AIN457 2x10mg/kg; AIN457 2x1.0mg/kg: AIN457A 1.0 mg/kg was administered intravenously as 2 doses 21 days apart, i.e. the first dose on day 1 and the second dose on day 22
- AIN457 2x0.1mg/kg: AIN457A 0.1 mg/kg was administered intravenously as 2 doses 21 days apart, i.e. the first dose on day 1 and the second dose on day 22
- Placebo: Placebo to AIN457A was administered intravenously as a single dose
Arm/Group | AIN457 2x10mg/kg | AIN457 2x1.0mg/kg | AIN457 2x0.1mg/kg | Placebo
Serious Adverse Events (participants affected / at risk) | 2/30 | 1/12 | 0/12 | 1/6
Other Adverse Events (participants affected / at risk) | 27/30 | 10/12 | 9/12 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AIN457 2x10mg/kg (N=30) | AIN457 2x1.0mg/kg (N=12) | AIN457 2x0.1mg/kg (N=12) | Placebo (N=6)
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 0 | 1 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AIN457 2x10mg/kg (N=30) | AIN457 2x1.0mg/kg (N=12) | AIN457 2x0.1mg/kg (N=12) | Placebo (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Cardiovascular insufficiency (Cardiac disorders) | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 2 | 1 | 0 | 1
Eye swelling (Eye disorders) | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 1 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 7 | 0 | 2 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Mouth ulceration (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 6 | 1 | 1 | 1
Oral mucosal eruption (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pancreatic enlargement (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Chills (General disorders) | 0 | 0 | 1 | 1
Fatigue (General disorders) | 3 | 0 | 3 | 1
Influenza like illness (General disorders) | 0 | 1 | 0 | 0
Malaise (General disorders) | 2 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 5 | 0 | 0 | 0
Temperature intolerance (General disorders) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 2 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 2 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 3 | 1 | 1 | 0
Nasopharyngitis (Infections and infestations) | 8 | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 2 | 1 | 0 | 0
Oral herpes (Infections and infestations) | 2 | 0 | 0 | 1
Otitis externa (Infections and infestations) | 2 | 0 | 0 | 0
Otitis media (Infections and infestations) | 1 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 2 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 1 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 1 | 0
Epicondylitis (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Aortic bruit (Investigations) | 0 | 0 | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Bone swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Tendon calcification (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Burning sensation (Nervous system disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 3 | 1 | 0 | 1
Dysaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 2 | 1 | 0 | 0
Headache (Nervous system disorders) | 7 | 1 | 3 | 0
Paraesthesia (Nervous system disorders) | 3 | 1 | 0 | 1
Sinus headache (Nervous system disorders) | 0 | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Dyshidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Circulatory collapse (Vascular disorders) | 2 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety